CLINICAL TRIAL: NCT02239484
Title: An Open-label, Randomized, Multiple-dose Crossover Study to Evaluate a Pharmacokinetic Drug Interaction Between Tadalafil and Tamsulosin in Healthy Male Volunteers
Brief Title: Evaluating a Pharmacokinetic Drug Interaction Between Tadalafil and Tamsulosin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM-TASU-101
Record Dates: First submitted 2014-09-04; First posted 2014-09-12 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Erectile Dysfunction; Benign Prostatic Hyperplasia
MeSH Terms: conditions — Erectile Dysfunction; Prostatic Hyperplasia | interventions — Tadalafil; Tamsulosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sequence 1 (Experimental): Tadalafil→Tamsulosin→Tadalafil+Tamsulosin
  Interventions: Drug: Tadalafil; Drug: Tamsulosin; Drug: Tadalafil + Tamsulosin
- Sequence 2 (Experimental): Tadalafil+Tamsulosin→Tadalafil→Tamsulosin
  Interventions: Drug: Tadalafil; Drug: Tamsulosin; Drug: Tadalafil + Tamsulosin
- Sequence 3 (Experimental): Tamsulosin→Tadalafil+Tamsulosin→Tadalafil
  Interventions: Drug: Tadalafil; Drug: Tamsulosin; Drug: Tadalafil + Tamsulosin

INTERVENTIONS:
Drug: Tadalafil
Drug: Tamsulosin
Drug: Tadalafil + Tamsulosin

SUMMARY:
We investigate the potential pharmacokinetic drug-drug interaction between Tadalafil and Tamsulosin in healthy male volunteers who receive Tadalafil alone, Tamsulosin alone, and both together in a 3 period repeatedly.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male volunteers, age 20 to 55 years.
2. The result of Body Mass Index(BMI) is not less than 19 kg/m2 , no more than 27 kg/m2
3. Subjects who have ability to comprehend the objectives, contents of study and property of study drug before participating in trial and have willingness to sign of informed consent in writing

Exclusion Criteria:

1. Presence of medical history or a concurrent disease that may interfere with treatment and safety assessment or completion of this clinical study, including clinically significant disorders in kidney, liver, cardiovascular system, respiratory system, endocrine system, or neuropsychiatric system.
2. Liver enzyme (AST, ALT) level exceeds one and a half times more than maximum normal range.
3. Systolic blood pressure <90mmHg or Diastolic blood pressure < 70 mmHg, systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg(Sitting blood pressure) during the screening procedure.

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Tadalafil,Tamsulosin Cmax,ss | 6day 0h(predose), 0.5, 1, 2, 3, 4, 6, 7, 8, 10, 12, 24, 48, 72 hours (Total 14)
Tadalafil,Tamsulosin AUCτ | 6day 0h(predose), 0.5, 1, 2, 3, 4, 6, 7, 8, 10, 12, 24, 48, 72 hours (Total 14)

SECONDARY OUTCOMES:
Tadalafil,Tamsulosin tmax,ss | 6day 0h(predose), 0.5, 1, 2, 3, 4, 6, 7, 8, 10, 12, 24, 48, 72 hours (Total 14)
Tadalafil,Tamsulosin t1/2 | 6day 0h(predose), 0.5, 1, 2, 3, 4, 6, 7, 8, 10, 12, 24, 48, 72 hours (Total 14)
Tadalafil,Tamsulosin CL/Fss | 6day 0h(predose), 0.5, 1, 2, 3, 4, 6, 7, 8, 10, 12, 24, 48, 72 hours (Total 14)
Tadalafil,Tamsulosin Vd/Fss | 6day 0h(predose), 0.5, 1, 2, 3, 4, 6, 7, 8, 10, 12, 24, 48, 72 hours (Total 14)
Tadalafil,Tamsulosin Cav | 6day 0h(predose), 0.5, 1, 2, 3, 4, 6, 7, 8, 10, 12, 24, 48, 72 hours (Total 14)
Tadalafil,Tamsulosin Cmin,ss | 6day 0h(predose), 0.5, 1, 2, 3, 4, 6, 7, 8, 10, 12, 24, 48, 72 hours (Total 14)

CONTACTS AND LOCATIONS:
Locations (1):
- Samgsung Seoul Hospital, Seoul, South Korea